CLINICAL TRIAL: NCT05588271
Title: Establishment of Risk Prediction Model for Pressure Injury in Patients Undergoing Liver Transplantation and Development of Prediction Tool
Brief Title: A New Prediction Mode for Predicting the Risk of Pressure Injury in Patients Undergoing Liver Transplantation
Acronym: PMPRPIULT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2022-178-B
Record Dates: First submitted 2022-10-18; First posted 2022-10-20 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Liver Transplantation
Keywords: Pressure injury; Liver transplantation; Predictive mode
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with PIs: stage 1pressure injury: non-blanchable erythema of intact skin; stage 2 pressure injury: partial-thickness skin loss with exposed dermis; stage 3 pressure injury: full-thickness skin loss; stage 4 pressure injury: full-thickness skin and tissue loss; unstageable pressure injury: obscured full-thickness skin and tissue loss; deep tissue pressure injury: persistent non-blanchable deep red, maroon or purple discoloration
  Interventions: Other: Exposures
- Group without PIs: Skin in good condition

INTERVENTIONS:
Other: Exposures — This study is an observational study.Exposure factors is patients with pressure injury.
  Groups: Group with PIs

SUMMARY:
Pediatric population is at a high-risk of pressure injury (PI). Patients undergoing liver transplantation are more prone to PIs compared with other types of surgery. However, there is a lack of sensitive and specific assessment tools for the risk of PI in patients undergoing liver transplantation. How to accurately predict the incidence of PI in patients undergoing liver transplantation is needs to be urgently eliminated. The study is conducted in the Renji Hospital, School of Medicine, Shanghai Jiaotong University which is the largest liver transplantation center in China.

DETAILED DESCRIPTION:
Data of 1200 eligible patients undergoing liver transplantation between July 2018 and June 2021 are selected.The sample size was randomly divided into 70% discovery set and 30% validation set according to 7:3. 70% of the discovery dataset are used for the establishment of risk prediction model. The univariate analysis is used to evaluate PI-associated risk factors. In addition, a multivariate logistic regression model is developed using selected variables and P<0.05 in the univariate analysis is used to identify independent risk factors for PIs. The odds ratio for each independent variable is determined with a 95% confidence interval. Finally, a nomogram of predictive model is generated on the basis of the results of multivariate analysis.Discrimination capability, calibration degree, and clinical value will be used to verify the efficacy of the prediction model. This study develops and validates a prediction model for predicting the risk of PI in patients undergoing liver transplantation. Using this prediction model, we will develop decision-support systems to prevent PI in the future.

ELIGIBILITY:
Inclusion Criteria:

* undergoing liver transplantation surgery (i.e., living-donor liver transplantation and deceased donor liver transplantation)
* patients undergoing the first surgery during their hospitalization

Exclusion Criteria:

* a history of PI before undergoing surgery
* patients with skin disease that could affect observation of skin and the outcome
* patients who died during surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing liver transplantation surgery
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
According to The National Pressure Ulcer Advisory Panel (NPUAP) defined the definition and stage of Pressure Injury to Judge whether pressure injury occurs on skin under pressure. | Within 6 hours after operation
  Definition:A pressure injury is localized damage to the skin and underlying soft tissue usually over a bony prominence or related to a medical or other device. The injury can present as intact skin or an open ulcer and may be painful. The injury occurs as a result of intense and/or prolonged pressure or pressure in combination with shear. The tolerance of soft tissue for pressure and shear may also be affected by microclimate, nutrition, perfusion, co-morbidities and condition of the soft tissue.
  NPUAP Pressure Injury Stages:stage 1pressure injury: non-blanchable erythema of intact skin; stage 2 pressure injury: partial-thickness skin loss with exposed dermis; stage 3 pressure injury: full-thickness skin loss; stage 4 pressure injury: full-thickness skin and tissue loss; unstageable pressure injury: obscured full-thickness skin and tissue loss; deep tissue pressure injury: persistent non-blanchable deep red, maroon or purple discoloration

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Chen, Master, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China